CLINICAL TRIAL: NCT04999462
Title: A Randomized, Parallel Trial to Assess the Effects of Replacing Non-fermented, Non-dairy Foods With Full-fat or Low-fat Fermented Dairy Foods on Insulin Sensitivity, RBC FA's and Other Markers of Cardiometabolic Health
Brief Title: A Trial to Assess Full-fat or Low-fat Dairy Foods on Insulin Sensitivity, RBC FA's and Other Markers of Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MB-1913
Record Dates: First submitted 2021-07-20; First posted 2021-08-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-09

CONDITIONS: Overweight and Obesity; Elevated Triglycerides
MeSH Terms: conditions — Overweight; Obesity; Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Full-fat fermented dairy (Experimental): 1 serving per day of full-fat yogurt and full-fat fermented cheese
  Interventions: Other: Full-fat fermented dairy
- Low-fat fermented dairy (Active Comparator): 1 serving per day of low-fat yogurt and lower-fat fermented cheese (e.g., reduced-fat or low-fat fermented cheese).
  Interventions: Other: Low-fat fermented dairy
- Non-dairy, non-fermented foods (Placebo Comparator): 2 servings per day of nondairy, nonfermented foods with a macronutrient composition that is similar to that of the low-fat fermented dairy condition.
  Interventions: Other: Non-dairy, non-fermented foods

INTERVENTIONS:
Other: Full-fat fermented dairy — Subjects assigned to the full-fat fermented dairy condition will consume 1 serving/d each of full-fat yogurt (plain or reduced sugar varieties) and full-fat fermented cheese.
  Arms: Full-fat fermented dairy
Other: Low-fat fermented dairy — Subjects assigned to the low-fat fermented dairy condition will consume 1 serving/d each of low-fat yogurt (plain or reduced sugar varieties) and lower-fat fermented cheese (e.g., reduced-fat or low-fat fermented cheese).
  Arms: Low-fat fermented dairy
Other: Non-dairy, non-fermented foods — Subjects assigned to the control condition will consume 2 servings/d of nondairy, nonfermented foods with a macronutrient composition that is similar to that of the low-fat fermented dairy condition.
  Arms: Non-dairy, non-fermented foods

SUMMARY:
The objectives of this trial are to assess the effects of adding 2 servings/d of either full-fat or low-fat fermented dairy products to the diet, as a replacement for non-dairy foods with macronutrient composition similar to the low-fat fermented dairy condition, on insulin sensitivity, erythrocyte fatty acid profile and other cardiometabolic health markers in metabolically at-risk adults.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18-74 years of age, inclusive.
2. Subject has a BMI of 25.00 kg/m2 to 39.99 kg/m2 at screening (visit 1b).
3. Subject has a fasting TG level ≥135 mg/dL at screening (visit 1a), or a fasting TG level 122-134 mg/dL (inclusive) and a fasting venous TG level of ≥135 mg/dL at screening (visits 1a and 1b, respectively).
4. Subject has a rating of 7 to 10 on the Vein Access Scale at screening (visit 1b; Appendix 2).
5. Subject is judged by the Investigator to be in general good health on the basis of medical history and screening laboratory tests.
6. Subject is willing to maintain usual physical activity pattern throughout the study and is willing to refrain from vigorous physical activity for 24 h prior to each clinic visit.
7. Subject has no plans to change smoking habits during the study and is willing to abstain from tobacco products and caffeine use 1 h prior to and during each clinic visit.
8. Subject is willing to refrain from using marijuana and consuming alcoholic beverages for 24 h prior to each clinic visit.
9. Subject is willing to consume study-related foods and follow the dietary instructions throughout the 12-week treatment period.
10. Subject is willing to come to the clinic for study food pick-up(s) if needed.
11. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator and is willing to complete study procedures.

Exclusion Criteria:

1. Subject has a laboratory test result of clinical significance at screening (visit 1b).
2. Subject has fasting blood glucose ≥126 mg/dL at screening (visit 1a) or known type 1 or type 2 diabetes mellitus.
3. Subject has atherosclerotic cardiovascular disease including any of the following: clinical signs of atherosclerosis including peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease [symptomatic (e.g., myocardial infarction, angina, transient ischemic attack or stroke of carotid origin) or >50% stenosis on angiography or ultrasound] or other forms of clinical atherosclerotic disease (e.g., renal artery disease).
4. Subject has a history or presence of a clinically important medical condition that, in the opinion of the investigator, could interfere with the interpretation of the study results.
5. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) at screening (visit 1b).
6. Subject has a history of cancer in the prior 5 years, except for non-melanoma skin cancer or carcinoma in situ of the cervix.
7. Subject has experienced a change in body weight of ±4.5 kg (10 pounds) over the 3 months prior to screening (visit 1b).
8. Subject has unstable use (initiation or dose alteration) of any antihypertensive medication within 4 weeks prior to screening (visit 1b).
9. Subject has unstable use (initiation or dose alteration) of any of the following lipid-altering medications within 4 weeks prior to screening (visit 1b): statins, ezetimibe, bempedoic acid, bile acid sequestrants, fibrates, niacin (drug form), and/or omega-3 fatty acid drugs.
10. Subject has unstable use (initiation or dose alteration) of a proprotein convertase subtilisin kexin type 9 (PCSK9) inhibitor within 3 months of screening (visit 1b).
11. Subject has unstable use (initiation or dose alteration) of weight-loss drugs (including over-the-counter medications and/or supplements) and/or systemic corticosteroid drugs within 4 weeks of screening (visit 1b).
12. Subject has unstable use (initiation or dose alteration) of medications known to influence carbohydrate metabolism, including, but not limited to: adrenergic receptor blockers, thiazide diuretics, hypoglycemic medications, and/or antipsychotics within 4 weeks prior to screening (visit 1b).
13. Subject has an active infection or has used antibiotics within 5 d of any clinic visit. Those with an active infection and/or using antibiotics must wait at least 5 d after the infection resolves or antibiotic use is complete. The test period will be extended for completion in these cases.
14. Subject has a known allergy, sensitivity, or intolerance to any ingredients in the study foods. Mild lactose intolerance is not exclusionary.
15. Subject is a female, who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
16. Subject has extreme dietary habits (e.g., vegan or very low carbohydrate diet).
17. Subject has a current or recent history (past 12 months), or strong potential, for drug or alcohol abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1 ½ oz distilled spirits).
18. Subject has a history of a diagnosed eating disorder (e.g., anorexia nervosa or bulimia nervosa).
19. Subject has been exposed to any non-registered drug product within 30 d of screening (visit 1b).
20. Subject has a condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 12 weeks
  The percent change from baseline to the end of treatment at 12 weeks in the Matsuda index

SECONDARY OUTCOMES:
Carbohydrate metabolism variables | 12 weeks
  Changes or percent changes from baseline to the end of treatment of fasting glucose and insulin, liquid meal tolerance test (LMTT) disposition index and homeostasis model assessments of pancreatic beta-cell function (HOMA2%B) and insulin sensitivity (HOMA2%S).
Lipid variables | 12 weeks
  Changes or percent changes from baseline to end of treatment of total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), non-high-density lipoprotein cholesterol (non-HDL-C), HDL-C, TG; lipoprotein particle concentrations and subfractions.
Erythrocyte | 12 weeks
  Changes or percent changes from baseline to the end of treatment of Erythrocyte 15:0, 17:0 and 1-16:1n-7 content (expressed as % of total fatty acids)
High-sensitivity C-reactive proten (hs-CRP) | 12 weeks
  Changes or percent changes from baseline to the end of treatment
Waist circumference | 12 weeks
  Changes or percent changes from baseline to the end of treatment
Seated, resting systolic and diastolic blood pressures and heart rate | 12 weeks
  Changes or percent changes from baseline to the end of treatment
Alternate Healthy Eating Index | 12 weeks
  Changes or percent changes from baseline to the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Study Director — MB Clinical Research & Consulting, LLC
Locations (4):
- United States (4):
  - Excellence Medical and Research, Miami Gardens, Florida
  - Illinois Institute of Technology, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Great Lakes Clinical Trials, Gurnee, Illinois

IPD SHARING:
Plan to Share IPD: No